CLINICAL TRIAL: NCT03833609
Title: Protocol for a Pilot Randomized Controlled Trial of the Evaluation of Yoga and Aerobic Dance for Pain Management in Juvenile Idiopathic Arthritis
Brief Title: Yoga and Aerobic Dance for Pain Management in Juvenile Idiopathic Arthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Children's Hospital of Eastern Ontario (Other)
Collaborators: The Hospital for Sick Children (Other); Université de Montréal (Other); University of Ottawa (Other)
Responsible Party: Principal Investigator, Karine Toupin-April, Associate Scientist, Children's Hospital of Eastern Ontario
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHEOREB#17/08X
Record Dates: First submitted 2018-11-26; First posted 2019-02-07 (Actual); Last update posted 2019-02-07 (Actual); Status verified 2019-02

CONDITIONS: Juvenile Idiopathic Arthritis; Pain
MeSH Terms: conditions — Arthritis, Juvenile; Pain

STUDY DESIGN:
Intervention Model Description: This study will use a three-arm prospective randomized open-label study. Participants will be randomized to one of the three following groups in a ratio of 2:2:1: A) an online yoga training program (+ physical activity (PA) electronic educational pamphlet) (n=10), B) an online aerobic dance training program (+ PA electronic educational pamphlet) (n=10) and C) a wait list control group (+ PA electronic educational pamphlet) (n=5). The total intervention period is 12 consecutive weeks. The frequency and duration of the intervention is based on other trials of yoga and physical activity interventions in pediatric and adult rheumatology.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Online yoga training (Group A) (Experimental): Participants will receive an e-pamphlet on physical exercise developed by The Arthritis Society, and will be invited to complete a yoga training program. The yoga training program is a structured low-intensity Vishwas-Raj. Participants will be asked to complete three individual 1-hour sessions per week for 12 consecutive weeks by watching a previously filmed session led by a qualified yoga instructor and posted on Facebook. They will also take part in a 1-hour virtual group session per week using a video-conferencing platform. Participants will also participate in weekly e-consultations with a research coordinator and discussions on Facebook with other participants.
  Interventions: Behavioral: Online yoga training (Group A)
- Online aerobic dance training (Group B) (Experimental): Participants will receive the e-pamphlet on physical exercise and will be invited to complete an aerobic dance program. The aerobic dance program is a low to moderate intensity level program and will also use a video. The video, adapted for youth with JIA, was developed with feedback from a JIA patient with experience in aerobic dance and a physiotherapist with experience in pediatric rheumatology. The aerobic dance program will have the same characteristics in terms of frequency, total number of sessions and total duration as the yoga program (i.e., three 1-hour individual sessions and one 1-hour virtual group session per week for 12 weeks). Participants will also participate in weekly e-consultations with a research coordinator and discussions on Facebook with other participants.
  Interventions: Behavioral: Online aerobic dance training (Group B)
- Wait list control (Group C) (No Intervention): Participants will receive the e-pamphlet on physical exercise and will be instructed to continue with their current medical care while they are on the wait list (12 weeks). After the completion of the study, the yoga and aerobic dance training videos will be available to all participants including those in the control group. In recruitment documents, this group will be termed the e-pamphlet group.

INTERVENTIONS:
Behavioral: Online yoga training (Group A) — The yoga training program is a structured low-intensity Vishwas-Raj (18). This yoga program consists of stretching, strengthening, meditation and deep breathing, and has been shown to be effective among adults with RA. Participants will be asked to complete three individual 1-hour sessions per week for 12 consecutive weeks by watching a previously filmed session led by a qualified yoga instructor and posted on Facebook. They will also take part in a 1-hour virtual group session per week using a video-conferencing platform. Participants will also participate in weekly e-consultations with a research coordinator and discussions on Facebook with other participants.
  Arms: Online yoga training (Group A)
Behavioral: Online aerobic dance training (Group B) — The aerobic dance program is a low to moderate intensity level program and will also use a video. The video, adapted for youth with JIA, was developed with feedback from a JIA patient with experience in aerobic dance and a physiotherapist with experience in pediatric rheumatology. The aerobic dance program will have the same characteristics in terms of frequency, total number of sessions and total duration as the yoga program (i.e., three 1-hour individual sessions and one 1-hour virtual group session per week for 12 weeks). Participants will also participate in weekly e-consultations with a research coordinator and discussions on Facebook with other participants.
  Arms: Online aerobic dance training (Group B)

SUMMARY:
The primary objectives of the proposed pilot randomized controlled trial (RCT) will be to examine: (1) the feasibility of a full RCT to evaluate the effectiveness of two popular types of physical activity (PA), a yoga training program and an aerobic dance training program, in female adolescents (13 to 18 years old) with juvenile idiopathic arthritis (JIA) compared to a wait list control group; and (2) the acceptability of these interventions. A three-arm prospective randomized open-label study with a parallel group design will be used. A total of 25 in a ratio of 2:2:1 female adolescents with JIA who have pain will be randomized to one of the three groups: 1) online yoga training program (Group A) (n=10), 2) online aerobic dance training program (Group B) (n=10) and 3) waiting list control group (Group C) (n=5). Participants in groups A and B will complete three individual 1-hour sessions per week using online exercise videos, as well as one 1-hour virtual group session per week using a video-conferencing platform (GoToMeeting) for 12 weeks. These participants will also take part in weekly e-consultations with a research coordinator and discussions on Facebook with other participants. Participants from all groups will be given access to an electronic educational pamphlet on PA for arthritis developed by The Arthritis Society to review via an online platform. Feasibility, acceptability and usability of Facebook and GoToMeeting will be assessed at the end of the program. Pain intensity (Primary outcome), participation in general physical activity, morning stiffness, functional status, fatigue, self-efficacy and patient global assessment will be assessed using self-administered electronic surveys at baseline, weekly until the end of the 12 weeks program.

DETAILED DESCRIPTION:
Objectives: The primary objectives of the proposed pilot randomized controlled trial (RCT) will be to examine: (1) the feasibility of a full RCT to evaluate the effectiveness of two popular types of physical activity (PA), a yoga training program and an aerobic dance training program, in female adolescents (13 to 18 years old) with juvenile idiopathic arthritis (JIA) compared to a wait list control group; and (2) the acceptability of these interventions.

Methods: A three-arm prospective randomized open-label study with a parallel group design will be used. A total of 25 female adolescents with JIA who have pain will be randomized in a ratio of 2:2:1 to one of the three groups: 1) online yoga training program (Group A) (n=10), 2) online aerobic dance training program (Group B) (n=10) and 3) wait list control group (Group C) (n=5). Participants in groups A and B will complete three individual 1-hour sessions per week using online exercise videos, as well as one 1-hour virtual group session per week using a video-conferencing platform (GoToMeeting) for 12 weeks. These participants will also take part in weekly e-consultations with a research coordinator and discussions on Facebook with other participants. Participants from all groups will be given access to an electronic educational pamphlet on PA for arthritis developed by The Arthritis Society to review via an online platform. Feasibility (recruitment rates, self-reported adherence to the interventions, dropout rates, and percentage of missing data), acceptability and usability of Facebook and GoToMeeting will be assessed at the end of the program. Pain intensity (Primary outcome), participation in general physical activity, morning stiffness, functional status, fatigue, self-efficacy and patient global assessment will be assessed using self-administered electronic surveys at baseline, weekly until the end of the 12 weeks program.

Conclusion: To our knowledge this is the first study in paediatric patients to evaluate the effectiveness of yoga and aerobic dance as pain management interventions for female adolescents with JIA. The use of online tools such as Facebook and GoToMeeting to disseminate these two PA interventions may facilitate access to alternative methods of pain management in this population. The study design incorporates randomization and allocation concealment to ensure internal validity. To avoid intergroup contamination, the Facebook group page security settings will be set to "closed", thus only allowing invited participants to access it. Study limitations include the lack of participant blinding due to the characteristics of this physical intervention pilot randomized controlled trial and a potential bias of recruiting more severe hospital-based participants. Reporting of the study follows the Standard Protocol Items: Recommendations for interventional trials (SPIRIT) statement. This study can lead to a full-scale RCT.

ELIGIBILITY:
Inclusion Criteria:

* Female adolescents aged between 13 -18 years old
* Diagnosis of JIA by a rheumatologist according to ILAR criteria
* Absence of serious co-morbidities, chronic diseases or of chronic pain that is unrelated to JIA (e.g., cancer, fibromyalgia), which may impact ability to understand and use the exercise program or complete outcome assessments (as determined by the treating rheumatologist)
* Presence of arthritis-related pain during regular activities of at least 30 on a 100-millimeter (mm) visual analogue scale (VAS) in the past month
* JIA specific medication regimen not expected to change during the study period
* Self-reported as not meeting Health Canada's and American College of Sports Medicine's guidelines for PA (<60 minutes of moderate to vigorous PA per day) and not using physical interventions/treatments other than medication prescribed for JIA pain relief or over the counter medication
* Capable of using and accessing the Internet weekly for the study duration
* No contraindications to exercise (according to the treating rheumatologist)
* Understand English

Exclusion Criteria:

* Moderate to severe cognitive impairments (as determined by the treating rheumatologist)
* Presence of serious co-morbidities, chronic illnesses or of chronic pain that is unrelated to JIA (e.g., cancer, fibromyalgia), which may impact ability to understand and use the exercise program or complete outcome assessments (as determined by the treating rheumatologist)
* Presence of pain during regular activities lower than 30mm on a 100 mm VAS in the past month
* Self-reported as physically active according to Health Canada's and American College of Sports Medicine's PA guidelines (≥60 minutes of moderate to vigorous PA per day) or using physical interventions/agents other than medication prescribed for JIA pain relief or over the counter medication
* JIA specific medication regimen expected to change during the study period
* Incapable of using and accessing the Internet weekly during the study duration
* Presence of contraindications to exercise
* Do not understand English

Ages: 13 Years to 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Estimated)
Dates: Start 2019-09 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate | This will be measured on a continued basis up to 12 weeks.
  The number of participants recruited in the trial and the time used for recruitment will be documented in a feasibility form. The number of participants will be divided by the time used for recruitment.
Randomization process | This will be measured on a continued basis up to 12 weeks.
  The ease at which the randomization process is conducted will be described by researchers in a feasibility form.
Number of protocol deviations | This will be measured on a continued basis up to 12 weeks.
  The number of protocol deviations, the time at which they occur, the group in which they occur and the potential reasons for these will be documented in a feasibility form. Participants will be asked the reasons why they deviated from the protocol by researchers using a feasibility form.
Dropout rates | This will be measured on a continued basis up to 12 weeks.
  The number of participants who drop out of the trial, the time at which they drop out, the group in which they belong and the reasons for these will be documented in a feasibility form. Participants will be asked the reasons why they drop out by researchers. The number of dropouts in each group will be divided by the time of the trial.
Percentage of missing data in the questionnaires | This will be measured on a continued basis up to 12 weeks.
  The percentage of missing data in the questionnaires, the time at which they occur and potential reasons for these will be documented in a feasibility form.
Self-reported adherence to the interventions using a modified Physical activity report calendar | This will be measured each week up to 12 weeks.
  Self-reported adherence to the aerobic dance and yoga training programs will be assessed by monitoring the number and length of sessions, and dividing the time spent performing the program by the time of prescribed sessions of either yoga or aerobic dance. Self-reported adherence will be recorded weekly using an adapted online version of the validated 7-day Physical Activity Report (PAR) calendar (in minutes).
Acceptability of the interventions: questionnaire | This will be assessed at 6 and 12 weeks.
  Acceptability of the yoga or aerobic dance interventions will be assessed using a questionnaire administered post-intervention. Questions will explore the acceptability of the e-consultations, virtual group sessions, the PA videos (either yoga or aerobic dance programs), the e-pamphlet and the training programs (content and duration of the yoga and aerobic dance programs), as well as facilitators and barriers to participating.
Usability of Facebook: System Usability Scale | This will be measured at 6 and 12 weeks.
  The usability of Facebook will be assessed by the System Usability Scale (SUS). The SUS is composed of 10 items using a 5-point scoring system ranging from Strongly disagree (score of 1 out of 5 for each question) to Strongly Agree (score of 5 out of 5 for each question). The total score ranges from 5 (low usability) to 50 (high usability).
Usability of GoToMeeting: System Usability Scale | This will be measured at 6 and 12 weeks.
  The usability of GoToMeeting will be assessed by the System Usability Scale (SUS). The SUS is composed of 10 items using a 5-point scoring system ranging from Strongly disagree (score of 1 out of 5 for each question) to Strongly Agree (score of 5 out of 5 for each question). The total score ranges from 5 (low usability) to 50 (high usability).
Use of Facebook | This will be measured at 6 and 12 weeks.
  The use of Facebook will be assessed by the number of posts, live online discussions and views of the videos.

SECONDARY OUTCOMES:
Change in pain intensity using the Childhood Health Assessment Questionnaire | This will be measured at baseline, 6 weeks and 12 weeks.
  Pain intensity will be assessed by the online Childhood Health Assessment Questionnaire (CHAQ) 100-mm pain VAS sub-scale. It uses a scoring system where 0 mm represents "no pain" and 100 mm "very severe pain" in the past week. This measure has already been validated in the JIA population. A repeated measures analysis of variance (ANOVA) with the fixed factor study group and the within factor assessment time (0, 6, 12 weeks) will be conducted to compare groups at 0, 6 and 12 weeks.
Change in level of physical activity using the Physical Activity Questionnaire for adolescents | This will be measured at baseline, 6 weeks and 12 weeks.
  Participation in physical activity will be assessed by the online Physical Activity Questionnaire for adolescents (PAQ-A) ages ranging from 14-18 years, a seven-day recall instrument measuring the level of physical activity within the last 7 days. The PAQ-A is composed of eight items using a 5-point scoring system. The total score is calculated by taking the mean score out of 5, with 1 indicating low physical activity and 5 indicating high physical activity. The PAQ-A has been reported to be a valid and reliable measure of general physical activity levels in youth and adolescents. A repeated measures analysis of variance (ANOVA) with the fixed factor study group and the within factor assessment time (0, 6, 12 weeks) will be conducted to compare groups at 0, 6 and 12 weeks.
Change in duration and intensity of physical activity using the Physical Activity Report Calendar | This will be measured at baseline, 6 weeks and 12 weeks.
  This will be assessed by an exercise log, based on the 7-day PAR calendar. Physical activity level will be reported in terms of minutes and intensity levels (three subscales: moderate, hard and very hard intensity: subscale total scores in minutes) and will be transformed into metabolic equivalent of tasks (METS), which are units of the basal metabolic rate and are expressing the energy cost of physical activity. A repeated measures analysis of variance (ANOVA) with the fixed factor study group and the within factor assessment time (0, 6, 12 weeks) will be conducted to compare groups at 0, 6 and 12 weeks.
Change in morning stiffness using self-reported questions | This will be measured at baseline, 6 weeks and 12 weeks.
  Morning stiffness will be assessed by online self-reported questions asking about the presence (Yes/No) and duration of morning stiffness in minutes. A repeated measures analysis of variance (ANOVA) with the fixed factor study group and the within factor assessment time (0, 6, 12 weeks) will be conducted to compare groups at 0, 6 and 12 weeks.
Change in functional status using the Childhood Health Assessment Questionnaire | This will be measured at baseline, 6 weeks and 12 weeks.
  Functional status will be assessed by the online Childhood Health Assessment Questionnaire (CHAQ). CHAQ contains 8 domains (dressing/grooming, arising, eating, walking, hygiene, reach, grip, and activities) and items are scored using a 4-point Likert scale of 0-3 where 0 represents the ability to perform the activity with no difficulty; 1, the ability to perform with some difficulty; 2, the ability to perform with much difficulty; and 3, the inability to perform over the past week. The mean of the 8 scores will determine the total CHAQ score ranging from 0 to 3, with a lower score indicating higher functional status and a higher score indicating lower functional status. It is the most widely used functional health status measure in JIA, which is a reliable and valid tool for the functional, physical and psychosocial assessment of children with JIA.
Change in fatigue using the PROMIS Pediatric Short Form v1.0 - Fatigue 10a | This will be measured at baseline, 6 weeks and 12 weeks.
  Fatigue will be assessed by an online version of a subset of the Patient-Reported Outcomes Measurement Information System (PROMIS) Pediatric Short Form v1.0 - Fatigue 10a which measures fatigue experiences and its impact, scored from 1 to 5, where 1 represents "never tired" and 5 "almost always tired" in the past week. A repeated measures analysis of variance (ANOVA) with the fixed factor study group and the within factor assessment time (0, 6, 12 weeks) will be conducted to compare groups at 0, 6 and 12 weeks.
Change in self-Efficacy using the Children's Arthritis Self-Efficacy Scale | This will be measured at baseline, 6 weeks and 12 weeks.
  Self-Efficacy will be assessed by the Children's Arthritis Self-Efficacy Scale (CASE), a specific valid and reliable tool for JIA. The CASE is an 11-item self-report scale that is divided into three concepts: activity, symptom and emotion. A 5-point Likert scale is used to rate responses for each item where 1 = "not at all sure" to 5 = "very sure" based on how confident the child is that they can manage disease effects. A repeated measures analysis of variance (ANOVA) with the fixed factor study group and the within factor assessment time (0, 6, 12 weeks) will be conducted to compare groups at 0, 6 and 12 weeks.
Patient Global Assessment using the Juvenile Arthritis Quality of Life Questionnaire | This will be measured at 6 weeks and 12 weeks.
  Patient Global Assessment will be assessed by an item used in the Juvenile Arthritis Quality of Life Questionnaire (JAQQ). The JAQQ was designed to assess the health-related quality of life in children aged 2-18 years with juvenile rheumatoid arthritis or juvenile spondylarthritides. The JAQQ includes four subscales (gross motor function, fine motor function, psychosocial function and systemic symptoms), as well as a pain and patient global assessment. The patient global assessment asks how youth have been since the last assessment (prior week) on a 5-point likert scale from much better (1) to much worse (5).

CONTACTS AND LOCATIONS:
Overall Officials: Karine Toupin April, Principal Investigator — Children's Hospital of Eastern Ontario
Locations (1):
- Children's Hospital of Eastern Ontario Research Institute, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No